CLINICAL TRIAL: NCT00003082
Title: A Phase IA Trial of Combined Murine IgG Monoclonal Anti-Transferrin Receptor Antibodies E2.3 and A27.15 in Cancer Patients
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Advanced Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Michael Lobell, M.D., Arizona Cancer Center at University of Arizona Health Science Center
Purpose: Treatment
Other Study IDs: CDR0000065781; P30CA023074 (NIH); UARIZ-HSC-95178; NCI-T96-0025
Record Dates: First submitted 1999-11-01; First posted 2004-07-19 (Estimated); Last update posted 2010-03-16 (Estimated); Status verified 2007-05

CONDITIONS: Chronic Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma and Plasma Cell Neoplasm; Myelodysplastic Syndromes; Precancerous/Nonmalignant Condition; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; monoclonal gammopathy of undetermined significance; recurrent adult Hodgkin lymphoma; isolated plasmacytoma of bone; extramedullary plasmacytoma; refractory multiple myeloma; Waldenstrom macroglobulinemia; stage III multiple myeloma; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; recurrent adult acute myeloid leukemia; recurrent adult acute lymphoblastic leukemia; relapsing chronic myelogenous leukemia; refractory chronic lymphocytic leukemia; unspecified adult solid tumor, protocol specific; chronic phase chronic myelogenous leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; adult acute myeloid leukemia in remission; adult acute lymphoblastic leukemia in remission; polycythemia vera; chronic idiopathic myelofibrosis; essential thrombocythemia; untreated hairy cell leukemia; progressive hairy cell leukemia, initial treatment; refractory hairy cell leukemia; chronic myelomonocytic leukemia; T-cell large granular lymphocyte leukemia; acute undifferentiated leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent adult Burkitt lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; recurrent adult T-cell leukemia/lymphoma; secondary acute myeloid leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; prolymphocytic leukemia; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; primary systemic amyloidosis; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; recurrent mantle cell lymphoma; angioimmunoblastic T-cell lymphoma; anaplastic large cell lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Myeloproliferative Disorders; Leukemia; Lymphoma; Multiple Myeloma; Neoplasms, Plasma Cell; Myelodysplastic Syndromes; Precancerous Conditions; Hodgkin Disease; Monoclonal Gammopathy of Undetermined Significance; Waldenstrom Macroglobulinemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Polycythemia Vera; Primary Myelofibrosis; Thrombocythemia, Essential; Leukemia, Hairy Cell; Leukemia, Myelomonocytic, Chronic; Leukemia, Large Granular Lymphocytic; Leukemia, Biphenotypic, Acute; Lymphoma, Follicular; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Burkitt Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Prolymphocytic; Immunoglobulin Light-chain Amyloidosis; Lymphoma, Mantle-Cell; Immunoblastic Lymphadenopathy; Lymphoma, Large-Cell, Anaplastic; Lymphoma, B-Cell, Marginal Zone

INTERVENTIONS:
Biological: monoclonal antibody A27.15
Biological: monoclonal antibody E2.3

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells.

PURPOSE: Phase I trial to study the effectiveness of monoclonal antibodies in treating patients who have advanced cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the toxicities associated with a 4-hour infusion of antitransferrin receptor antibodies with one antibody administered by itself for 1 hour before the second antibody infusion is started. II. Determine the pharmacokinetics of monoclonal antibodies E2.3 and A27.15.

OUTLINE: This is a dose escalating study. Patients receive antitransferrin antibody A27.15 IV over 4 hours. One hour after the initiation of the A27.15 infusion, infusion of antibody E2-3 is added by IV piggy back. In the absence of antimouse antibodies and toxic effects, treatment continues once every 4 weeks in patients achieving minimal, partial, or complete remission. Treatment ceases in patients experiencing stable or progressive disease. In the absence of dose limiting toxicity in the first 3 patients treated, subsequent cohorts of 6 patients each receive escalating doses of antitransferrin antibodies E2.3 and A27.15 on the same dose schedule. If dose limiting toxicity occurs in 2 of 6 patients at a given dose level, then dose escalation ceases and the next lower dose is declared the MTD. Patients are followed for 3 weeks.

PROJECTED ACCRUAL: This study will accrue 18-27 patients within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Refractory or recurrent advanced malignancy following known standard effective therapy or advanced malignancy for which no standard effective therapy exists Measurable or evaluable disease

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: SWOG 0-2 Life expectancy: At least 2 months Hematopoietic: Absolute neutrophil count at least 1800/mm3 Hematocrit at least 30 mg/dL Platelet count at least 50,000/mm3 Hepatic: Bilirubin no greater than 1.5 times normal unless due to disease, then less than 3.5 times normal Transaminases less than 3 times upper limit of normal (ULN) (less than 5 times ULN if due to liver metastases) Renal: Creatinine no greater than 2.5 times normal Cardiovascular: No severe cardiac abnormalities Must have adequate venous access No history of sustained ventricular arrhythmia or unexplained syncope Pulmonary: No severe pulmonary abnormalities Other: Not pregnant or nursing Effective contraception required of fertile female patients No serious concurrent medical or psychiatric illness Adequate nutrition No human antimouse antibodies

PRIOR CONCURRENT THERAPY: At least 4 weeks since prior anticancer therapy and recovered If there was disease progression during therapy, at least 2 weeks since prior anticancer therapy and recovered Biologic therapy: Not specified Chemotherapy: No concurrent chemotherapy Endocrine therapy: Concurrent topical steroids used in the chronic management of cutaneous T cell lymphoma allowed No other concurrent hormone therapy Radiotherapy: No concurrent palliative radiotherapy Surgery: Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Estimated)
Dates: Start 1997-12; Primary Completion 2001-02 (Actual); Study Completion 2001-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lobell, MD, Study Chair — University of Arizona
Locations (1):
- Arizona Cancer Center, Tucson, Arizona, United States